CLINICAL TRIAL: NCT01578343
Title: A Phase II Investigation of Vorinostat in Combination With Intravenous Fludarabine, Mitoxantrone, and Dexamethasone in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Vorinostat Plus FND in Relapsed or Refractory Mantle Cell Lymphoma
Acronym: ZOLINZA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: we collected data of a total of 19 patients for an interim analysis. but there are less than 7 responses out of the initial 19 patients.
Sponsor: Samsung Medical Center (Other)
Collaborators: Seok Jin Kim (Unknown)
Responsible Party: Principal Investigator, Won Seog Kim, Associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC2011-11-102-001
Record Dates: First submitted 2012-03-30; First posted 2012-04-16 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: fludarabine; mitoxantrone; dexamethasone; relapsed or refractory mantle cell lymphoma; FND regimen; vorinostat; autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — fludarabine; Mitoxantrone; Dexamethasone; Vorinostat; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat-FND (Experimental): Vorinostat-fludarabine, mitoxantrone, dexamethasone Induction treatment (Total 4 cycles) FND D1-3 Fludarabine 25mg/m2 + NS 100mL iv over 30 min D1 Mitoxantrone 10mg/m2 + NS 100mL iv over 30 min D1-5 Dexamethasone 20mg IV or PO every 4 weeks Vorinostat D1-10 Vorinostat 200mg once daily PO (When vorinostat is concurrently administered with FND regimen, vorinostat will be administered 3 hours before chemotherapy)
  Interventions: Drug: Fludarabine, Mitoxantrone, Dexamethasone, Vorinostat

INTERVENTIONS:
Drug: Fludarabine, Mitoxantrone, Dexamethasone, Vorinostat — 1. Induction treatment (Total 4 cycles) FND D1-3 Fludarabine 25mg/m2 + NS 100mL iv over 30 min D1 Mitoxantrone 10mg/m2 + NS 100mL iv over 30 min D1-5 Dexamethasone 20mg IV or PO every 4 weeks Vorinostat D1-10 Vorinostat 200mg once daily PO (When vorinostat is concurrently administered with FND regimen, vorinostat will be administered 3 hours before chemotherapy)
  2. Consolidation treatment for responders Patients not eligible for transplantation
     * Vorinostat maintenance up to 6 cycles
     * 200mg twice daily for 14 consecutive days from D1 - 14 in a 21 day cycle
     * Delay of the start of the next cycle by up to 7 days will be acceptable.
     * If relapse or progression during maintenance, it will be stopped. Patients eligible for transplantation
     * High-dose chemotherapy followed by autologous stem cell transplantation
  Other Names: 1.Induction treatment (Total 4 cycles) D1-3 Fludarabine D1 Mitoxantrone D1-5 Dexamethasone Vorinostat D1-10 Vorinostat; 2.Consolidation treatment for responders Patients not eligible for transplantation

SUMMARY:
1. Rationale In mantle cell lymphoma, the conventional chemotherapy achieves only temporary responses with a median duration of remissions only from 1 to 2 years. Therefore, mantle cell lymphoma is known as one of the B-cell lymphomas with poor prognosis. Although the treatment outcome of mantle cell lymphoma has been improved since intensive chemotherapy regimens such as HyperCVAD was used, a substantial number of patients are still frequently relapsed after chemotherapy. After relapse, most of them became refractory to various kinds of salvage treatment. That is why the results of most salvage chemotherapy regimens were disappointing. In addition, mantle cell lymphoma generally occurs in elderly people. Thus, intensive salvage chemotherapy may not be feasible for elderly patients. Therefore, an effective, novel combination treatment is urgently needed in relapsed or refractory mantle cell lymphoma patients.
2. Hypothesis

   * Vorinostat will produce synergism with a combination treatment regimen (Fludarabine, mitoxantrone, dexamethasone, FND) without overlapping toxicity
   * Vorinostat maintenance treatment will reduce the relapse rate in patients ineligible for autologous stem cell transplantation.
3. Purpose A phase II investigation to determin the effectiveness of vorinostat in combination with intravenous fludarabine, mitoxantrone, and dexamethasone in patients with relapsed or refractory mantle cell lymphomain patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
1. Objectives 1.1 Primary objective • To determine the efficacy of vorinostat plus FND as an induction treatment

   * Response rate of vorinostat/FND 1.2 Secondary objective

     * Survival outcome
   * Overall survival and progression-free survival

     * To determine the efficacy of vorinostat maintenance treatment
   * Relapse rate • Toxicity of vorinostat/FND
   * Hematologic and non-hematologic toxicity

ELIGIBILITY:
1. Inclusion

   * Histologically proven mantle cell lymphoma
   * Adequate organ function as defined by the following criteria:

     * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
     * Total serum bilirubin ≤1.5 x ULN
     * Absolute neutrophil count (ANC) ≥1500/µL
     * Platelets ≥100,000/µL
     * Hemoglobin ≥9.0 g/dL (may be transfused or erythropoietin treated)
     * Serum calcium ≤12.0 mg/dL
     * Serum creatinine ≤1.5 x ULN
     * Normal potassium and magnesium at baseline
   * All patients should be relapsed or refractory patients after previous treatments including chemotherapy .
   * At least one measurable lesion (lymph node or tumor mass)

     - The size of lesion must be > 1.0cm in the greatest transverse diameter
   * ECOG PS 0-2
   * Serum HCG test: negative if a patient is female eligible for pregnancy
2. Exclusion

   * Major surgery or radiation therapy within 4 weeks of starting the study treatment.
   * History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease or secondary CNS involvement on CT or MRI scan.
   * Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
   * Pregnancy or breastfeeding.
   * Patients with HIV positive
   * Patients with HBs antigen positive
   * Patients with anti-HCV positive
   * History of the use of another HDAC inhibitor: e.g. valproic acid

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of vorinostat plus FND as an induction treatment confirmed by CT or MRI (PET/CT as indicated) | A) After 8weeks and 16 weeks of the treatment
  B) Response criteria
  1) Complete response (CR): Disappearance of all detectable clinical and radiographic evidence of disease 2) Partial response (PR): ≥50% decrease in sum of product diameter (SPD) of 6 nodes/nodal masses 3) Stable disease (SD): Disease status is less than PR, but is not PD 4) Progressive disease (PD): Appearance of any new lesions

SECONDARY OUTCOMES:
To determine the efficacy of vorinostat maintenance treatment, survival outcome and toxicity of vorinostat/FND measured by CT or MRI scan, CTCAE ver 4.0 | every 3 months during the 1st two years after enrollment
  A) Disease status evaluation every 3 months during the 1st two years after enrollment B) Monitoring survival status during the five years after enrollment C) Toxicity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Meical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
we will share collected data with principal investigator in Korea